CLINICAL TRIAL: NCT03095573
Title: Prospective Randomized Comparison Between Axial- and Lateral-viewing Capsule Endoscopy Systems in Celiac Patients: a Pilot Study
Brief Title: Comparison Between Axial- and Lateral-viewing Capsule Endoscopy in Celiac Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Collaborators: IRCCS Policlinico S. Donato (Other)
Responsible Party: Principal Investigator, Luca Elli, MD, PhD, Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: Capsocam
Record Dates: First submitted 2017-03-20; First posted 2017-03-29 (Actual); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Celiac Disease
Keywords: Celiac disease; Enteropathy associated T cell lymphoma; Refractory celiac disease; Small bowel adenocarcinoma
MeSH Terms: conditions — Celiac Disease; Enteropathy-Associated T-Cell Lymphoma

STUDY DESIGN:
Intervention Model Description: Each enrolled patients will undergo examination of the small bowel by means of both endoscopic capsule devices (the axial-view PillCam SB3 and the lateral-view CapsoCam) on the same day at approximately 3 hours interval from one another. The order of administration of the two different capsules will be determined by a specific randomization sequence.
Who Masked: Outcomes Assessor
Masking Description: The videos will be reviewed by three experts operators blinded about the sequence of capsule examination administration
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Lateral-viewing capsule (Experimental): Examination of the small bowel by means of the lateral-viewing CapsoCam device
  Interventions: Device: Lateral-viewing CapsoCam device
- Axial-viewing capsule (Active Comparator): Examination of the small bowel by means of the axial-viewing capsule
  Interventions: Device: Axial-viewing capsule

INTERVENTIONS:
Device: Lateral-viewing CapsoCam device — Small bowel capsule endoscopy examination with the Lateral-viewing CapsoCam device
  Arms: Lateral-viewing capsule
Device: Axial-viewing capsule — Small bowel capsule endoscopy examination with the Axial-viewing capsule device
  Arms: Axial-viewing capsule

SUMMARY:
Video capsule endoscopy (VCE) is recommended as the gold standard in small bowel exploration. The efficiency of the axial-viewing (Given, Imaging) has been widely reported. The CapsoCam capsule (Capsovision, California, USA) has four cameras allowing the exploration of the small bowel through 360 degree lateral viewing. Celiac disease is the most common autoimmune enteropathy in Western countries, and is usually associated with a good response to the gluten free diet and an excellent prognosis. However, a minority of patients develop complications of the disease, such as refractory celiac disease, ulcerative jejunoileitis and neoplastic complications such as adenocarcinoma of the small bowel and enteropathy associated T cell lymphoma. In recent years, the detection of small bowel lesions has dramatically improved thank to the availability of capsule endoscopy exploration. The aim of this study was to evaluate detection rate and diagnostic concordance of the axial view capsule and CapsoCam capsules in the same patients.

DETAILED DESCRIPTION:
The study will involve 25 patients with suspected complicated celiac disease , which for clinical reasons are referred for an evaluation of the small intestine by means of capsule endoscopic in order to screen/identify complications. Furthermore, patients under regular follow-up for a known complication of celiac disease (i.e. refractory celiac disease, ulcerative jejunoileitis) will also be enrolled.

Patients reffered to the Center for Prevention and Diagnosis of celiac disease at the research Hospital "Fondazione Cà Granda Ospedale Maggiore Policlinico" in Milan will be prospectively evaluated and consecutively enrolled in the study.

In agreement with international Guidelines, the diagnosis of celiac disease will be based on Presence of atrophy in the duodenal biopsy sampling (Marsh-Oberhuber type 3) and positive serology or genetic compatibility (in case of seronegative patients at diagnosis).

Patients at high risk of celiac disease complications are defined as

* subjects older than 50 years at the time of celiac disease diagnosis
* subjects with persistence / recurrence of gastrointestinal symptoms after at least 6 months of gluten-free diet
* subjects reporting poor compliance to the gluten-free diet
* subjects with alarm signs at diagnosis or during follow-up.

All enrolled patients will undergo examination of the small bowel by means of both endoscopic capsule devices (the axial-view PillCam SB3 and the lateral-view CapsoCam) on the same day at approximately 3 hours interval from one another, according to a protocol already validated in terms of security in other studies. The order of administration of the two different capsules, will be determined by a specific randomization sequence.

At the end of the examination, recorded data from the capsules will be acquired according to the following steps:

* For the axial-view capsule: removal of the recorder after 10 hours recording and/or after checking that the capsule has reached the cecum. The patient will also be instructed to retrieve the capsule from the stools in the hours / days following the examination as per standard protocol.
* For the lateral-view capsule, the patient will be given a specific kit for its retrieval and conservation. The recorded data will be downloaded after retrieval of the capsule.

The 50 videos will be reviewed by three experts operators (L.E., F.B. G.E.T.), blinded and in randomized order. The operators will evaluate the number of lesions detected by the two different types of capsule system (Primary endpoint) and the mean extension of the lesions detected, expressed as percentage of the total transit time of the capsule in the small intestine (Secondary endpoint)

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with celiac disease at high risk of complication (see above for a detailed description)

Exclusion Criteria:

* presence of Pacemaker or Defibrillator
* suspected small bowel obstruction
* impaired swallowing
* pregnancy
* presence of contraindications to a capsule endoscopy examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-10-31 (Estimated); Study Completion 2019-02-28 (Estimated)

PRIMARY OUTCOMES:
Lesions detected | up to 24 hours, the time of progression of the capsule through the small bowel
  Mean number of lesions detected by the two different types of devices, expressed as diagnostic yield and total number of lesions

SECONDARY OUTCOMES:
Extension of the lesions | up to 24 hours, the time of progression of the capsule through the small bowel
  Mean extension of the lesions detected, expressed as percentage of the total transit time of the capsule in the small intestine

CONTACTS AND LOCATIONS:
Overall Officials: Luca Elli, MD, PhD, Principal Investigator — Fondazione IRCCS Ca´Granda Ospedale Maggiore Policlinico, Milano, Italy
Locations (2):
- Italy (2):
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan, MI
  - Irccs Policlinico San Donato, San Donato Milanese, MI

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Volta U, Bellentani S, Bianchi FB, Brandi G, De Franceschi L, Miglioli L, Granito A, Balli F, Tiribelli C. High prevalence of celiac disease in Italian general population. Dig Dis Sci. 2001 Jul;46(7):1500-5. doi: 10.1023/a:1010648122797. PMID 11478502
- [Background] Green PH, Fleischauer AT, Bhagat G, Goyal R, Jabri B, Neugut AI. Risk of malignancy in patients with celiac disease. Am J Med. 2003 Aug 15;115(3):191-5. doi: 10.1016/s0002-9343(03)00302-4. PMID 12935825
- [Background] Catassi C, Bearzi I, Holmes GK. Association of celiac disease and intestinal lymphomas and other cancers. Gastroenterology. 2005 Apr;128(4 Suppl 1):S79-86. doi: 10.1053/j.gastro.2005.02.027. PMID 15825131
- [Background] Culliford A, Daly J, Diamond B, Rubin M, Green PH. The value of wireless capsule endoscopy in patients with complicated celiac disease. Gastrointest Endosc. 2005 Jul;62(1):55-61. doi: 10.1016/s0016-5107(05)01566-x. PMID 15990820
- [Background] Daum S, Wahnschaffe U, Glasenapp R, Borchert M, Ullrich R, Zeitz M, Faiss S. Capsule endoscopy in refractory celiac disease. Endoscopy. 2007 May;39(5):455-8. doi: 10.1055/s-2007-966239. PMID 17516353
- [Background] Rondonotti E, Spada C, Cave D, Pennazio M, Riccioni ME, De Vitis I, Schneider D, Sprujevnik T, Villa F, Langelier J, Arrigoni A, Costamagna G, de Franchis R. Video capsule enteroscopy in the diagnosis of celiac disease: a multicenter study. Am J Gastroenterol. 2007 Aug;102(8):1624-31. doi: 10.1111/j.1572-0241.2007.01238.x. Epub 2007 Apr 24. PMID 17459022
- [Background] Rostom A, Murray JA, Kagnoff MF. American Gastroenterological Association (AGA) Institute technical review on the diagnosis and management of celiac disease. Gastroenterology. 2006 Dec;131(6):1981-2002. doi: 10.1053/j.gastro.2006.10.004. No abstract available. PMID 17087937
- [Background] Rondonotti E, Soncini M, Girelli C, Ballardini G, Bianchi G, Brunati S, Centenara L, Cesari P, Cortelezzi C, Curioni S, Gozzini C, Gullotta R, Lazzaroni M, Maino M, Mandelli G, Mantovani N, Morandi E, Pansoni C, Piubello W, Putignano R, Schalling R, Tatarella M, Villa F, Vitagliano P, Russo A, Conte D, Masci E, de Franchis R; AIGO, SIED and SIGE Lombardia. Small bowel capsule endoscopy in clinical practice: a multicenter 7-year survey. Eur J Gastroenterol Hepatol. 2010 Nov;22(11):1380-6. doi: 10.1097/MEG.0b013e3283352ced. PMID 20173646
- [Background] Bardella MT, Elli L, De Matteis S, Floriani I, Torri V, Piodi L. Autoimmune disorders in patients affected by celiac sprue and inflammatory bowel disease. Ann Med. 2009;41(2):139-43. doi: 10.1080/07853890802378817. PMID 18777226
- [Background] Leighton JA. The role of endoscopic imaging of the small bowel in clinical practice. Am J Gastroenterol. 2011 Jan;106(1):27-36; quiz 37. doi: 10.1038/ajg.2010.410. Epub 2010 Oct 26. PMID 20978483
- [Background] Pioche M, Vanbiervliet G, Jacob P, Duburque C, Gincul R, Filoche B, Daudet J, Filippi J, Saurin JC; French Society of Digestive Endoscopy (SFED). Prospective randomized comparison between axial- and lateral-viewing capsule endoscopy systems in patients with obscure digestive bleeding. Endoscopy. 2014 Jun;46(6):479-84. doi: 10.1055/s-0033-1358832. Epub 2013 Nov 27. PMID 24285122